CLINICAL TRIAL: NCT03965819
Title: A Randomized, Double-blind, Placebo-controlled, Cross-over, Pilot Study to Investigate the Efficacy of Pain Bloc-R in Healthy Participants With Non-pathological Aches and Discomfort
Brief Title: A Study to Investigate the Efficacy of Pain Bloc-R in Healthy Participants With Non-pathological Aches and Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeSeasons Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 18PPHL
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: Aches; Discomfort; Healthy; Adults; Body aches
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, cross-over
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All products look identical in identical opaque capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Randomized to consume Pain Bloc-R, Acetaminophen, then placebo (Experimental): Each study product will be consumed as 2 capsules daily for 7 days. Randomized to consume Investigational Natural Health Product in Study Period 1, Comparator in Study Period 2, and Placebo in Study Period 3.
  Interventions: Dietary Supplement: Pain Bloc-R; Other: Active Comparator - Acetaminophen; Other: Placebo
- Randomized to consume Acetaminophen, Placebo, then Pain Bloc-R (Experimental): Each study product will be consumed as 2 capsules daily for 7 days. Randomized to consume Comparator in Study Period 1, Placebo in Study Period 2, and the Investigational Product in Study Period 3.
  Interventions: Dietary Supplement: Pain Bloc-R; Other: Active Comparator - Acetaminophen; Other: Placebo
- Randomized to consume Placebo, Pain Bloc-R, then Acetaminophen (Experimental): Each study product will be consumed as 2 capsules daily for 7 days. Randomized to consume Placebo in Study Period 1, Investigational Product in Study Period 2, and Comparator in Study Period 3.
  Interventions: Dietary Supplement: Pain Bloc-R; Other: Active Comparator - Acetaminophen; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Pain Bloc-R — Herbal Supplement containing Vit D3, Vit B6, Vit B12, White Willow Bark, Angelica Root, Acetyl L-carnitine HCl, Caffeine, L-Theanine, Benfotiamine, and L-Tetrahydropalmatine
Other: Active Comparator - Acetaminophen — DIN 02447479 Encapsulated for Blinding Purposes
Other: Placebo — No active ingredients

SUMMARY:
A randomized, double-blind, placebo-controlled, cross-over pilot study to investigate the efficacy of Pain Bloc-R in healthy participants with non-pathological aches and discomfort. The study will have 3 study periods. During each study period, eligible participants will consume either Pain Bloc-R, comparator product, or placebo for 7 days during each study period (1 product per study period), with a 1-week washout period in between each period. The primary objective is the comparison of change in unresolved aches and discomfort from pre-supplement to Day 7 between the Pain Bloc-R, comparator, and placebo, as assessed by the Brief Pain Inventory (BPI) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18-65 years of age, inclusive
2. BMI of 18-32.5 kg/m2, inclusive
3. Individuals with occupational (construction workers, manual labourers, athletes) and non-occupational unresolved aches and discomfort for at least 2 weeks
4. Individuals on non-prescription, OTC medication for unresolved aches and discomfort and are willing to undergo a washout determined by the QI based on dose and frequency prior to enrollment
5. Female participants not of child bearing potential, defined as females who have had a hysterectomy or bilateral oophorectomy, bilateral tubal ligation, total endometrial ablation or are post-menopausal (natural or surgically with > 1 year since last menstruation) or, Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
6. Healthy as determined by laboratory results and medical history as assessed by the QI
7. Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits
8. Agrees to comply with study procedures
9. Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the trial
2. Anticipated problems or allergy to any ingredients in the investigational products
3. Allergy to rescue medication
4. Have chronic disease conditions causing chronic pain
5. Uncontrolled high and low blood pressure
6. Uncontrolled blood sugar levels
7. Clinically significant abnormal laboratory results at screening
8. Prescribed medications used to help with aches and discomfort (Section 7.3.1)
9. OTC medications and supplements taken to help with aches and discomfort (Section 7.3.2)
10. Autoimmune disease or if immune-compromised (i.e. HIV-positive, use of anti-rejection medication, rheumatoid arthritis, Hepatitis B/C-positive)
11. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow-up that is negative. Volunteers with cancer in full remission for more than 5 years after diagnosis are acceptable after review by QI
12. History of mental illness that might impair the ability of participants to provide written informed consent
13. Current or history of bleeding disorders
14. Current or history of liver or kidney disease as assessed by QI on a case by case basis.
15. Current or pre-existing unstable thyroid condition. Treatment on a stable dose medication for over one year will be reviewed on a case-by-base basis by the QI
16. Surgical procedures which may impact the study outcomes within the past 3 months to be assessed by the QI
17. Medicinal marijuana
18. Recreational marijuana; dose and frequency to be assessed by QI
19. Alcohol intake >2 standard drinks per day or >10 standard drinks per week
20. Illicit drug use in the past 6 months as assessed by the QI
21. Participation in clinical trials within 30 days prior to screening visit
22. Blood donation during or within 30 days after conclusion of clinical trial
23. Any other active or unstable medical condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Comparison of change in unresolved aches and discomfort from pre-supplementation to Day 7 between Pain Bloc-R, comparator and placebo as assessed by the Brief Pain Inventory (BPI) questionnaire | 7 days
  The Brief Pain Inventory (BPI) questionnaire developed by MD Anderson Cancer Centre is a discomfort assessment tool used to score an individual's level of discomfort severity and discomfort interference.
  Part A of the questionnaire evaluates pain severity, asking the participants to rate their "worst", "least", "average" and "right now" (current) levels of pain on a scale of 0 (no pain) to 10 (as bad as you can imagine).
  Part B evaluates the pain interference levels, asking the participants to rate the impact of their pain on their general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. Together, part A and part B aim to serve as a concise quantification tool for the pain levels and the participant's resulting quality of life. The questionnaire will be administered at each visit to monitor changes in participant's pain over the course of each phase.

SECONDARY OUTCOMES:
Comparison between Pain Bloc-R formula, comparator, and placebo in the change in musculoskeletal discomfort (MD) from pre-supplementation to Day 7 post-supplementation as assessed by modified Cornell musculoskeletal discomfort questionnaire | 7 days
  The modified Cornell Musculoskeletal Discomfort Questionnaire (mCMDQ) tool is used to assess physical discomfort. The questionnaire includes a list of body parts with an image for visualization. The questionnaire assesses the discomfort frequency score, from "never" (Rating Score = 0), "1-2 times/week" (RS 1.5), "3-4 times/week" (RS 3.5), "every day" (RS 5) and "several times a day" (RS 10). The questionnaire assesses discomfort severity score, as "slightly uncomfortable" (RS 1), "moderately uncomfortable" (RS = 2) or "very uncomfortable" (RS 3). Finally, the questionnaire determines the discomfort interference score, as "not at all" (RS 1), "slightly interfered" (RS 2), or "interfered a lot" (RS 3). The total discomfort score is calculated by multiplying the individual frequency, severity and interference scores for each body part, and then summed to yield a total discomfort score.
Comparison between Pain Bloc-R formula, comparator, and placebo in the change in general discomfort from pre-supplementation to Day 7 post-supplementation as assessed by the BPI questionnaire | 7 days
  The Brief Pain Inventory (BPI) questionnaire developed by MD Anderson Cancer Centre is a discomfort assessment tool used to score an individual's level of discomfort severity and discomfort interference.
  Part A of the questionnaire evaluates pain severity, asking the participants to rate their "worst", "least", "average" and "right now" (current) levels of pain on a scale of 0 (no pain) to 10 (as bad as you can imagine).
  Part B evaluates the pain interference levels, asking the participants to rate the impact of their pain on their general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. Together, part A and part B aim to serve as a concise quantification tool for the pain levels and the participant's resulting quality of life. The questionnaire will be administered at each visit to monitor changes in participant's pain over the course of each phase.
Comparison between Pain Bloc-R formula, comparator, and placebo in the proportion of participants consuming rescue medicine when taking Pain Bloc-R, comparator, or placebo | 7 days
Comparison between Pain Bloc-R formula, comparator, and placebo in Product perception and tolerability as assessed by the product perception questionnaire | 7 days
  A questionnaire containing 7 questions regarding the participants satisfaction, tolerability, and feelings toward the study product. The product perception questionnaire will be scored from 5,4,3,2,1 for strongly agree, agree, no opinion, disagree, strongly disagree respectively on each question. Min and max scores for each question are 1 and 5. The total score of the 7 questions is the sum scores of each question with the min and max of 1 and 35. The higher score indicates better product perception for each question and total score.

OTHER OUTCOMES:
The incidence of pre- and post-emergent adverse events (AEs) in the Pain Bloc-R formula, comparator, and placebo groups from pre-supplementation to Day 7 | 7 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on systolic blood pressure from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on diastolic blood pressure from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on heart rate from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on weight from pre-supplementation to Day 7 post-supplementation | 7 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on body mass index (BMI) from pre-supplementation to Day 7 post-supplementation | 7 days
  Weight and Height are measured. BMI is calculated by kg/m2.
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on clinical chemistry from screening to end-of-study as assessed by alanine aminotransferase (ALT) levels in the blood | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on clinical chemistry from screening to end-of-study as assessed by aspartate aminotransferase (AST) levels in the blood | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on clinical chemistry from screening to end-of-study as assessed by bilirubin levels in the blood | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on clinical chemistry from screening to end-of-study as assessed by creatinine levels in the blood | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on clinical chemistry from screening to end-of-study as assessed by sodium levels in the blood | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on clinical chemistry from screening to end-of-study as assessed by potassium levels in the blood | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on clinical chemistry from screening to end-of-study as assessed by chloride levels in the blood | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on hematology from screening to end-of-study as assessed by hemoglobin | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on hematology from screening to end-of-study as assessed by hematocrit | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on hematology from screening to end-of-study as assessed by platelet count | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on hematology from screening to end-of-study as assessed by red blood cell (RBC) count | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on hematology from screening to end-of-study as assessed by red blood cell (RBC) indices | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on hematology from screening to end-of-study as assessed by red cell distribution width (RDW) | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on hematology from screening to end-of-study as assessed by white blood cell (WBC) count | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on hematology from screening to end-of-study as assessed by neutrophils | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on hematology from screening to end-of-study as assessed by lymphocytes | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on hematology from screening to end-of-study as assessed by monocytes | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on hematology from screening to end-of-study as assessed by eosinophils | Between 42-87 days
The effect of supplementation with Pain Bloc-R formula, comparator, or placebo on hematology from screening to end-of-study as assessed by basophils | Between 42-87 days

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — Qualified Investigator
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No